CLINICAL TRIAL: NCT04180540
Title: A Randomized Comparison of Percutaneous Closure to Manual Compression for Hemostasis of Multiple Venous Access Sites Among Patients Undergoing Catheter Ablation for Atrial Fibrillation
Brief Title: Comparison of Percutaneous Closure to Manual Compression for Hemostasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael S. Lloyd (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor-Investigator, Michael S. Lloyd, Associate Professor, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00115958
Record Dates: First submitted 2019-11-26; First posted 2019-11-27 (Actual); Results first posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Atrial Fibrillation
Keywords: Cardiology; Electrophysiology
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Percutaneous Closure (Experimental): Participants randomized to undergo percutaneous closure with PerClose after radiofrequency ablation or cryoablation for treatment of atrial fibrillation.
  Interventions: Device: Percutaneous Closure
- Manual Compression (Active Comparator): Participants randomized to undergo manual compression after radiofrequency ablation or cryoablation for treatment of atrial fibrillation.
  Interventions: Other: Manual Compression

INTERVENTIONS:
Device: Percutaneous Closure — The PerClose Proglide system will be used to deliver a suture to close the venous puncture following completion of ablation for treatment of atrial fibrillation.
  Other Names: PerClose Proglide
  Arms: Percutaneous Closure
Other: Manual Compression — Manual compression is the standard method of attaining hemostasis following ablation for treatment of atrial fibrillation. Manual compression may be performed with or without "figure of eight" suture for hemostasis at the discretion of the treating physician).
  Arms: Manual Compression

SUMMARY:
This a prospective randomized trial occurring in patients undergoing routine ablation for atrial fibrillation as standard of care. The purpose of this study is to determine if using a small internal suture (or "stitch") facilitates faster times to hemostasis (stopping bleeding) after removing intravenous sheaths (special IVs that are used for ablation procedures) after an atrial fibrillation ablation procedure. The device used to place the stitch is PerClose Proglide and is an already FDA-approved technology for closing these IV sites. The study will also determine if it is safe to get up and walk sooner than what is considered typical after closing these IV sites with the PerClose device. Participants will be randomized in a 1:1 ratio to either manual compression or use of the PerClose for hemostasis at the end of the ablation procedure. The length of follow-up will be up to 30 days at routine clinical follow-up after the procedure.

DETAILED DESCRIPTION:
Radiofrequency ablation and cryoablation for treatment of atrial fibrillation (AF) using percutaneous venous access at the groin is one of the most common procedures performed by cardiac electrophysiologists. However, compared to other catheter-based interventions, patients undergoing AF ablation pose a unique set of challenges. First, AF ablation requires multiple points of transfemoral venous access with large diameter sheaths, ranging in size from 8 French gauge (F) to 14F for cryoablation procedures. Second, operators are forced to balance the competing risk of thrombosis and bleeding in these patients. In order to minimize the risk of intraprocedural thrombosis, anticoagulation with heparin with a goal anticoagulation time (ACT) >300-350 seconds is necessary. However, operators typically require ACTs to normalize prior to removal of sheaths and manual compression, which significantly delays hemostasis and ambulation. While reversal agents are an option, there is currently clinical equipoise on their role and safety in this setting and they require additional time to exert their full effect. Lastly, patients require at least 1-2 months of therapeutic oral anticoagulation after the procedure to mitigate ongoing stroke risk. These factors culminate in longer times to hemostasis and ambulation and raise concerns for post-procedure access related complications for patients undergoing AF ablation. PerClose Proglide has recently gained FDA approval for closure of percutaneous venous access sites for catheter-based interventions and remains the only commercially available solution for access sites >14F inner diameter. Percutaneous closure of venotomy sites may facilitate rapid hemostasis without the need for reversal of anticoagulation, potentially attenuating bleeding risk. Additionally, typical bedrest times after percutaneous closure are based on data derived from arterial closure. Prior limited data, as well as frequent anecdotal reports, have suggested that earlier ambulation may be feasible. Because the venous circulation is a lower pressure system, it is possible that earlier than standard ambulation times after PerClose is both safe and feasible. However, a rigorous prospective investigation of the PerClose Proglide device in the context of AF ablation has not been performed.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective atrial fibrillation ablation at Emory University Hospital or Emory University Hospital Midtown

Exclusion Criteria:

* women who are pregnant (based on standard pre-procedure pregnancy test)
* patients who are not able to ambulate pre-procedure
* patients who are unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lloyd, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory Clinic, Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Percutaneous Closure | Manual Compression
Started | 55 | 54
Completed | 53 | 54
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Percutaneous Closure | Manual Compression | Total
Number analyzed (Participants) | 55 | 54 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (10.0) | 64.3 (11.5) | 62.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 39 | 36 | 75
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 49 | 48 | 97
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 54 | 54 | 108
Baseline anticoagulation [Count of Participants; unit: Participants]
  Aspirin | 10 | 9 | 19
  Clopidogrel/P2Y12 inhibitor | 1 | 0 | 1
  Warfarin | 4 | 3 | 7
  Rivaroxaban | 8 | 10 | 18
  Dabigatran | 1 | 0 | 1
  Apixaban | 36 | 35 | 71
  None | 3 | 5 | 8
Medical History [Count of Participants; unit: Participants]
  Hypercholesterolemia | 17 | 20 | 37
  Hypertension | 33 | 30 | 63
  Peripheral Vascular Disease | 3 | 2 | 5
  Deep Vein Thrombosis | 0 | 1 | 1
  Cerebrovascular Disease | 2 | 3 | 5
  Congestive Heart Failure | 7 | 5 | 12
  Coronary Artery Disease | 6 | 13 | 19
  Prior groin access procedure | 18 | 21 | 39
  Current or ex-smoker | 19 | 14 | 33
  Diabetes | 6 | 5 | 11
  Cancer | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Time to Hemostasis
Description: Starting from sheath pull, time (in minutes) to hemostasis will be compared between study arms.
Time Frame: Day 1
Measure: Mean (Full Range); unit: seconds
Arm/Group | Percutaneous Closure | Manual Compression
Number analyzed (Participants) | 53 | 54
seconds | 4.5 [1.0 to 11.6] | 10.7 [9.7 to 14.2]

2. Secondary Outcome: Time to Ambulation
Description: Time to ambulation (in minutes) following the atrial fibrillation ablation, will be compared between study arms.
Time Frame: Day 1
Population: Of those in the Percutaneous Closure group (n=53), two patients were excluded as they had crossed over to full MC, and 5 others did not undergo secondary randomization due to lack of research staff or logistic challenges. Secondary randomization for six others was deferred at the discretion of the treating provider. Number of those who underwent secondary randomization (n=40).
Measure: Mean (Full Range); unit: Hours
Arm/Group | Percutaneous Closure | Manual Compression
Number analyzed (Participants) | 40 | 54
Hours | 1.33 [1.23 to 2.50] | 2.25 [1.91 to 3.20]

3. Secondary Outcome: Number of Complications
Description: Number of complications will be compared between study arms as a composite of all major access site complications and venous thromboembolism.
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Closure | Manual Compression
Number analyzed (Participants) | 53 | 54
Participants
  Complications at Discharge | 0 | 1
  Complications At follow Up | 0 | 1

4. Secondary Outcome: Short-form Inguinal Pain Questionnaire Score
Description: The Short-form Inguinal Pain Questionnaire is a quality of life metric where respondents report how much pain they have experienced in the past week and how pain has limited their activities. The questionnaire consists of two items, each with a score ranging from 0 to 6. Question 1 asks participants to report the worst pain they have experienced in the past week, where responses range from 0 (no pain) to 6 (pain present, prompt medical advice sought). If participants have experienced pain, Question 2 asks what limitations the pain has caused in performing everyday activities such as sitting down, standing up, or exercising. The total score for question 2 ranges from 0 (none of the listed activities were impacted) to 6 (all listed activities were impacted).
Time Frame: Day 30
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Percutaneous Closure | Manual Compression
Number analyzed (Participants) | 53 | 54
score on a scale
  Worst pain felt in the groin over the past 7 days | 0 [0 to 0] | 0 [0 to 0]
  Extent of limitation of ability to perform different activities by groin pain | 0 [0 to 0] | 0 [0 to 0]

5. Secondary Outcome: Procedure Length
Description: The length of the procedure to reach hemostasis, in minutes, will be compared between study arms.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Percutaneous Closure | Manual Compression
Number analyzed (Participants) | 53 | 54
minutes
  Initial Stick to Out of Lab | 158.06 (35.653) | 156.83 (54.346)
  Initial Stick to complete hemostasis | 141.81 (35.401) | 146.15 (53.805)

6. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction was assessed with a 6-item instrument where participants responded on a scale from 0 to 5 where 0 = completely satisfied and 5 = completely dissatisfied. The sum of scores can range from 0 to 30 and lower scores indicate greater satisfaction with pain level and appearance of the access site. Measurements were taken at discharge (day 1) and the same instrument was used on follow up (day 30).
Time Frame: Day 1 and Day 30
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Percutaneous Closure | Manual Compression
Number analyzed (Participants) | 53 | 54
score on a scale
  Pain in your Groin at Discharge | 1.13 (1.455) | 0.72 (1.14)
  Pain in your Groin at Day 30 | 0.59 (1.206) | 0.25 (0.845)
  Tenderness around your groin at Discharge | 1.21 (1.405) | 0.65 (1.067)
  Tenderness around your groin at Day 30 | 0.84 (1.546) | 0.49 (1.084)
  Numbness in your groin area at Discharge | 0.42 (0.719) | 0.3 (0.743)
  Numbness in your groin area at Day 30 | 0.29 (0.764) | 0.08 (0.392)
  Bruising around your groin area at Discharge | 0.7 (1.249) | 0.52 (1.077)
  Bruising around your groin area at Day 30 | 0.73 (1.44) | 0.84 (1.488)
  Problems in your groin where the catheter was inserted at Discharge | 0.49 (0.869) | 0.37 (0.938)
  Problems in your groin where the catheter was inserted at Day 30 | 0.29 (0.913) | 0.37 (0.937)
  Appearance of your bruise at Discharge | 0.64 (1.128) | 0.41 (0.962)
  Appearance of your bruise at Day 30 | 0.8 (1.581) | 0.92 (1.719)
  Sum of Scores | 4.58 (4.99) | 2.96 (4.813)

7. Secondary Outcome: Pain Medication Needs
Description: Post-procedure narcotic usage for pain medication requirements after hemostasis until discharge from the post-procedure area will be compared between study arms.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Closure | Manual Compression
Number analyzed (Participants) | 53 | 54
Participants | 8 | 5

8. Secondary Outcome: Costs
Description: Overall costs (in dollars) related to hemostasis and any complications over 30 days will be compared between study arms.
Time Frame: Day 30
Measure: Median (Inter-Quartile Range); unit: dollars
Arm/Group | Percutaneous Closure | Manual Compression
Number analyzed (Participants) | 53 | 54
dollars
  Cost related to Hemostasis | 882 [747 to 1,176] | 4 [4 to 163]
  Total cost of procedure | 882 [814.5 to 1,176] | 42 [4 to 163]
  Total cost of care related to procedure | 57,050.44 [47,251.40 to 66,426.34] | 56,533.65 [45,699.47 to 66,987.64]

9. Secondary Outcome: Number of Nursing Encounters
Description: The number of nursing encounters while in the post-procedure area will be compared between study arms.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: Number of encounters
Arm/Group | Percutaneous Closure | Manual Compression
Number analyzed (Participants) | 53 | 54
Number of encounters | 0.06 (0.231) | 0.09 (0.564)

ADVERSE EVENTS:
Time Frame: Event data was collected from baseline during procedure, to follow up 30 days after baseline
Arm/Group | Percutaneous Closure | Manual Compression
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/54
Serious Adverse Events (participants affected / at risk) | 2/53 | 1/54
Other Adverse Events (participants affected / at risk) | 4/53 | 12/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Percutaneous Closure (N=53) | Manual Compression (N=54)
Hematoma at Discharge (Cardiac disorders) | 2 (2) | 0 (0) — Hematoma on Closure at time of Discharge
Hematoma at Follow up (Cardiac disorders) | 0/51 (0) | 1/53 (1) — Hematomas assessed on Follow up visit
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Percutaneous Closure (N=53) | Manual Compression (N=54)
Minor Hematoma at Discharge (Cardiac disorders) | 1/51 (1) | 1 (1) — Minor Hematoma assessed at time of discharge
Minor Rebleeding or Ooze at Discharge (Cardiac disorders) | 3/51 (3) | 10 (10) — Minor Rebleeding or oozing assessed at time of discharge
Minor Hematoma at Follow Up (Cardiac disorders) | 0/51 (0) | 2/53 (2) — Minor Hematoma assessed at follow up visit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT04180540/Prot_000.pdf
  • Informed Consent Form (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT04180540/ICF_001.pdf